CLINICAL TRIAL: NCT04368988
Title: A 2-Part, Phase 1/2, Randomized, Observer-Blinded Study To Evaluate The Safety And Immunogenicity Of A SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine (SARS-CoV-2 rS) With Or Without MATRIX-M™ Adjuvant In Healthy Subjects
Brief Title: Evaluation of the Safety and Immunogenicity of a SARS-CoV-2 rS Nanoparticle Vaccine With/Without Matrix-M Adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-101
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Placebo - Phase 1 (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 1
- SARS-CoV-2 rS - 25 μg without Matrix-M - Phase 1 (Experimental): 2 doses of SARS-CoV-2 rS - 25 μg, 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS - Phase 1
- SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M - Phase 1 (Experimental): 2 doses of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (mixed together for each injection), 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 1
- SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M - Phase 1 (Experimental): 2 doses of SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M (mixed together for each injection), 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 1
- SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M then Placebo - Phase 1 (Experimental): 1 dose of SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M (mixed together for injection), on Day 0 followed by 1 dose of Placebo on Day 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M Adjuvant, Day 0 - Phase 1; Other: Normal saline solution (NSS), Placebo, Day 21 - Phase 1
- Placebo - Phase 2 (Placebo Comparator): 3 doses of Placebo (Saline), 1 dose each on Days 0, 21, and 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2
- SARS-CoV-2 rS - 5/5 μg + 50 μg Matrix-M - Phase 2 (Experimental): 2 doses of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (co-formulated), 1 dose each on Days 0 and 21, followed by 1 dose of Placebo on Day 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2; Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2
- SARS-CoV-2 rS - Alternating 5/5 μg + 50 μg Matrix-M - Phase 2 (Experimental): 1 dose of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (co-formulated) on Day 0 then 1 dose of Placebo on Day 21 followed by 1 dose of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (co-formulated) on Day 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2; Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2
- SARS-CoV-2 rS - 25/25 μg + 50 μg Matrix-M - Phase 2 (Experimental): 2 doses of SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M (co-formulated), 1 dose each on Days 0 and 21, followed by 1 dose of Placebo on Day 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2; Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2
- SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M - Phase 2 (Experimental): 1 dose of SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M (co-formulated) on Day 0 then 2 doses of Placebo, 1 dose each on Days 21 and 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2; Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2
- SARS-CoV-2 rS - 5/5/5 μg + 50 μg Matrix-M - Phase 2 (Experimental): 3 doses of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (co-formulated), 1 dose each on Day 0, Day 21, and Day 189.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2
- SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M - Phase 2 (Experimental): 1 dose of SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M (co-formulated) on Day 0 then 2 doses of Placebo, 1 dose each on Days 21 and 189.
  Interventions: Other: Normal saline solution (NSS), Placebo - Phase 2; Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2

INTERVENTIONS:
Biological: SARS-CoV-2 rS - Phase 1 — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS (0.6 mL) on Days 0 and 21.
  Arms: SARS-CoV-2 rS - 25 μg without Matrix-M - Phase 1
Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 1 — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS mixed with Matrix-M adjuvant (0.6 mL) on Days 0 and 21.
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M - Phase 1; SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M - Phase 1
Other: Normal saline solution (NSS), Placebo - Phase 1 — Alternating intramuscular (deltoid) injections of placebo (0.6 mL) on Days 0 and 21.
  Other Names: Sodium chloride solution for injection, 0.9%
  Arms: Placebo - Phase 1
Other: Normal saline solution (NSS), Placebo - Phase 2 — Intramuscular (deltoid) injections of placebo (0.5 mL).
  Other Names: Sodium chloride solution for injection, 0.9%
  Arms: Placebo - Phase 2; SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 25/25 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 5/5 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - Alternating 5/5 μg + 50 μg Matrix-M - Phase 2
Biological: SARS-CoV-2 rS/Matrix-M Adjuvant, Day 0 - Phase 1 — Intramuscular (deltoid) injection of SARS-CoV-2 rS mixed with Matrix-M adjuvant (0.6 mL) on Day 0.
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M then Placebo - Phase 1
Other: Normal saline solution (NSS), Placebo, Day 21 - Phase 1 — Intramuscular injection of placebo (0.6 mL) in alternate deltoid on Day 21.
  Other Names: Sodium chloride solution for injection, 0.9%
  Arms: SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M then Placebo - Phase 1
Biological: SARS-CoV-2 rS/Matrix-M Adjuvant - Phase 2 — Intramuscular (deltoid) injections of SARS-CoV-2 rS co-formulated with Matrix-M adjuvant (0.5 mL).
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS - 25 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 25/25 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 5 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 5/5 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - 5/5/5 μg + 50 μg Matrix-M - Phase 2; SARS-CoV-2 rS - Alternating 5/5 μg + 50 μg Matrix-M - Phase 2

SUMMARY:
2019nCoV-101 is a 2-part, randomized, observer-blinded, placebo-controlled, Phase 1/2 trial. Part 1 (Phase 1) of the study is designed to evaluate the safety and immunogenicity of SARS-CoV-2 rS nanoparticle vaccine with or without Matrix-M adjuvant in 131 healthy participants ≥ 18 to 59 (inclusive) years of age at 2 sites in Australia. An interim analysis of Part 1 safety and immunogenicity will be performed prior to optional expansion to Part 2. Part 2 (Phase 2) of the study is designed to evaluate the immunogenicity, safety, and preliminary efficacy of a single construct of SARS-CoV-2 rS nanoparticle vaccine with Matrix-M adjuvant in up to 1,500 healthy participants ≥ 18 to 84 (inclusive) years of age at up to 40 sites across Australia and/or the United States.

ELIGIBILITY:
Inclusion Criteria (Part 1):

* Healthy adult males or females between 18 and 59 years of age, inclusive, at screening. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
* The participant has a body mass index 17 to 35 kg/m2, inclusive, at screening.
* Willing and able to give informed consent prior to study enrollment and comply with study procedures.
* Female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months or documented plasma follicle-stimulating hormone (FSH) level ≥40 mIU/mL]) must agree to be heterosexually inactive from at least 21 days prior to enrollment and through 6 months after the last vaccination OR agree to consistently use any of the described methods of contraception from at least 21 days prior to enrollment and through 6 months after the last vaccination.

Exclusion Criteria (Part 1):

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care, inclusive of changes in medication in the past 2 months indicating that chronic illness/disease is not stable (at the discretion of the investigator). This includes any current workup of undiagnosed illness that could lead to a new condition.
* Chronic disease inclusive of: a) hypertension uncontrolled for age according to the Eighth Joint National Committee (JNC 8) guidelines; b) congestive heart failure by New York Heart Association (NYHA) functional classification of greater or equal to II; c) chronic obstructive pulmonary disease by Global Initiative for Obstructive Lung Disease (GOLD) classification of greater or equal to 2; d) recent (within 6 months prior to first study vaccination) exacerbation of coronary artery disease as manifested by cardiac intervention, addition of new cardiac medications for control of symptoms, or unstable angina; e) asthma (diagnosed by spirometry showing reversibility of disease and must meet at least the Step 1 classification with current prescription/use of medications to control symptoms); f) diabetes requiring use of medicine (insulin or oral) or not controlled with diet.
* Participation in research involving an investigational product (drug/biologic/device) within 45 days prior to first study vaccination.
* History of a confirmed diagnosis of SARS or COVID-19 disease (confirmed by a specific test for each disease) or known exposure to a SARS-CoV-2 positive confirmed close contact (eg, family member, housemate, daycare provider, aged parent requiring care), at the discretion of the investigator.
* Currently working in an occupation with a high risk of exposure to SARS-CoV-2 (eg, healthcare worker, emergency response personnel).
* Currently taking any product (investigational or off-label) for prevention of COVID-19 disease.
* Positive rapid test for SARS-CoV-2 (either ELISA IgG or PCR) at screening or prior to first vaccination. Testing may be repeated during the screening period if exposure to SARS-CoV-2 is suspected, at the discretion of the investigator.
* Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 4 weeks prior to first study vaccination.
* Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital).
* Chronic administration (defined as more than 14 continuous days) of immunosuppressant, systemic glucocorticosteroids, or other immune-modifying drugs within 90 days prior to first study vaccination; or anticipation of the need for immunosuppressive treatment within 6 months after last vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination.
* Any acute illness concurrent or within 14 days prior to first study vaccination (medical history and/or physical examination) or documented temperature of >38°C during this period. This includes respiratory or constitutional symptoms consistent with SARS-CoV-2 (COVID-19) exposure (ie, cough, sore throat, difficulty breathing).
* Known disturbance of coagulation (iatrogenic or congenital).
* Evidence of Hepatitis B or C or HIV by laboratory testing.
* A positive test result for drugs of abuse (except a positive test result associated with prescription medication that has been reviewed and approved by the investigator) or alcohol at screening.
* Any neurological disease or history of significant neurological disorder (eg, meningitis, seizures, multiple sclerosis, vasculitis, migraines, Guillain-Barré syndrome [genetic/congenital or acquired]).
* Active cancer (malignancy) within 5 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma, at the discretion of the investigator)
* Vital sign (blood pressure, pulse, temperature) abnormalities of toxicity grade >1.
* Clinical laboratory abnormalities of toxicity grade >1 for selected serum chemistry and hematology parameters
* Any known allergies to products contained in the investigational product or latex allergy.
* Women who are pregnant, breastfeeding or who plan to become pregnant during the study.
* History of alcohol abuse or drug addiction within 1 year prior to the first study vaccination.
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
* Study team member or first-degree relative of any study team member (inclusive of sponsor, PPD, and site personnel involved in the study).

Inclusion Criteria (Part 2):

* Healthy adult males or females between 18 and 84 years of age, inclusive, at screening who are of legal adult age in their local jurisdiction. Healthy status will be determined by the investigator based on medical history, clinical laboratory results, vital sign measurements, and physical examination at screening.
* The participant has a body mass index 17 to 35 kg/m2, inclusive, at screening.
* Willing and able to give informed consent prior to study enrollment and comply with study procedures.
* Female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months or documented plasma FSH level ≥40 mIU/mL]) must agree to be heterosexually inactive from at least 21 days prior to enrollment and through 6 months after the last vaccination OR agree to consistently use any of the following methods of contraception from at least 21 days prior to enrollment and through 6 months after the last vaccination.

Exclusion Criteria (Part 2):

* Participants who are having any current workup of undiagnosed illness within the last 8 weeks, which is either participant-reported or has been clinician-assessed, that could lead to a new condition diagnosis.
* Participation in research involving an investigational product (drug/biologic/device) within 45 days prior to first study vaccination.
* History of a confirmed diagnosis of SARS or history of a confirmed diagnosis of COVID-19 disease resulting in medical intervention.
* Received influenza vaccination within 14 days prior to first study vaccination, or any other vaccine within 4 weeks prior to first study vaccination.
* Have clinically significant chronic cardiovascular, endocrine, gastrointestinal/ hepatic, renal, neurological, respiratory, or other medical disorders not excluded by other exclusion criteria, that are assessed by the Investigator as being clinically unstable within the prior 4 weeks evidenced by: a) hospitalization for the condition, including day surgical interventions, b) new significant organ function deterioration, c) needing addition of new treatments or major dose adjustments of current treatments.
* Diabetes mellitus requiring insulin therapy (either type 1 or type 2 diabetes mellitus).
* Chronic obstructive pulmonary disease with a history of an acute exacerbation of any severity in the prior year.
* Any history of congestive heart failure.
* Any history of chronic kidney disease (the presence of impaired or reduced kidney function lasting at least 3 months). Clinical validation of potential cases of chronic kidney disease should be conducted.
* Evidence of unstable coronary artery disease as manifested by cardiac intervention, addition of new cardiac medications for control of symptoms, or unstable angina in the past 3 months.
* History of chronic neurological disorders that have required prior specialist physician review for diagnosis and management (such as multiple sclerosis, dementia, transient ischemic attacks, Parkinson's disease, degenerative neurological conditions, neuropathy, and epilepsy) or a history of stroke or previous neurological disorder within 12 months with residual symptoms. Participants with a history of migraine or chronic headaches or nerve root compression that have been stable on treatment for the last 4 weeks are not excluded.
* Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital).
* Chronic administration (defined as more than 14 continuous days) of immunosuppressants, systemic glucocorticosteroids reaching an immunosuppressive dose, or other immune-modifying drugs within 90 days prior to first study vaccination.
* Received immunoglobulin, blood-derived products, or other immunosuppressant drugs within 90 days prior to first study vaccination.
* Known disturbance of coagulation (iatrogenic or congenital).
* Active cancer (malignancy) within 5 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma, at the discretion of the investigator).
* Any known allergies to products contained in the investigational product or latex allergy.
* Women who are breastfeeding or who plan to become pregnant during the study.
* History of alcohol abuse or drug addiction within one year prior to the first study vaccination.
* Any condition that, in the opinion of the investigator, would pose a health risk to the subject if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
* Study team member or first-degree relative of any study team member (inclusive of sponsor, PPD, and site personnel involved in the study).

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1419 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Participants with Solicited Adverse Events (AEs) - Phase 1 | 28 days
  Percentage of participants with solicited AEs (local, systemic) for 7 days following each primary vaccination (Days 0, 21) by severity score, duration, and peak intensity.
Safety Laboratory Values (Serum Chemistry, Hematology) - Phase 1 | 28 days
  Safety laboratory values (serum chemistry, hematology) by FDA toxicity scoring (absolute and change from baseline where identified) at 7 days after each vaccination.
Serum Immunoglobulin G (IgG) Antibody Levels Expressed as Geometric Mean Titers (GMTs) - Phase 1 | 21 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMTs through Day 21.
Serum Immunoglobulin G (IgG) Antibody Levels Expressed as Geometric Mean Titers (GMTs) - Phase 1 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMTs through Day 35.
Serum IgG Antibody Levels Expressed as Geometric Mean Fold Rises (GMFRs) - Phase 1 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs through Day 35.
Serum IgG Antibody Levels Expressed as Seroconversion Rates (SCRs) - Phase 1 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs through Day 35. SCR is the proportion of participants with ≥4-fold rises in ELISA units.
Serum IgG Antibody Levels Expressed as GMEUs - Phase 2 | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs for the two-dose regimens by dose at Day 35 regardless of baseline immune status and stratified by baseline immune status.
Serum IgG Antibody Levels Expressed as GMFRs - Phase 2 | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs for the two-dose regimens by dose at Day 35 regardless of baseline immune status and stratified by baseline immune status.
Serum IgG Antibody Levels Expressed as SCRs - Phase 2 | Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs (≥4-fold rises) for the two-dose regimens by dose at Day 35 regardless of baseline immune status and stratified by baseline immune status.
Participants with Solicited Adverse Events (AEs) - Phase 2 | 28 days
  Percentage of participants with solicited AEs (local, systemic) for 7 days following each primary vaccination (Days 0 and 21) by severity score, duration, and peak intensity.
Participants with Unsolicited AEs - Phase 2 | 35 days
  Percentage of participants with unsolicited AEs (eg, treatment-emergent, serious, suspected unexpected serious, those of special interest, all medically attended adverse events [MAAEs]) through the 35 days by Medical Dictionary of Regulatory Activities (MedDRA) classification, severity score, and relatedness.

SECONDARY OUTCOMES:
Participants with Unsolicited AEs - Phase 1 | 49 days
  Percentage of participants with unsolicited AEs (eg, treatment-emergent, serious, suspected unexpected serious, those of special interest, all MAAEs) through the first 49 days by MedDRA classification, severity score, and relatedness.
Participants with Abnormal Vital Signs - Phase 1 | 21 days
  Percentage of participants with vital sign abnormalities on the day of vaccination by severity scoring immediately following vaccination.
Changes from Baseline in Body Temperature - Phase 1 | 189 days
  Mean changes from baseline in body temperature by treatment group and visit.
Changes from Baseline in Blood Pressure - Phase 1 | 189 days
  Mean changes from baseline in blood pressure by treatment group and visit.
Changes from Baseline in Pulse Rate - Phase 1 | 189 days
  Mean changes from baseline in pulse rate by treatment group and visit.
Participants with MAAEs - Phase 1 | 105 days
  Percentage of participants with MAAEs, defined as AEs that lead to an unscheduled visit to a healthcare practitioner, through Day 105 by MedDRA classification, severity score, and relatedness.
Participants with Related MAAEs; Serious Adverse Events (SAEs); and Adverse Events of Special Interest (AESI) - Phase 1 | 386 days
  Percentage of participants with MAAEs assessed as related to study vaccine, SAEs, and AESIs until the end of the study (EOS) by MedDRA classification and severity score. All SAEs and AESI, defined as potential immune-mediated medical conditions or AEs relevant to COVID-19, by MedDRA classification, severity score, and relatedness.
Assessment of Serum IgG Antibody Levels Expressed as GMTs at Multiple Time Points - Phase 1 | 189 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at multiple time points through Day 189.
Assessment of Serum IgG Antibody Levels Expressed as GMFRs at Multiple Time Points - Phase 1 | 189 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at multiple time points through Day 189.
Assessment of Serum IgG Antibody Levels Expressed as SCRs at Multiple Time Points - Phase 1 | 189 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs (proportion of participants with ≥2-fold and ≥4-fold rises in antibody levels) at multiple time points through Day 189.
Assessment of Serum IgG Antibody Levels Expressed by Seroresponse Rates (SRRs) at Multiple Time Points - Phase 1 | 189 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SRRs (proportion of participants with rises in ELISA units exceeding the 95th percentile of placebo participants) at multiple time points through Day 189.
Angiotensin-Converting Enzyme 2 (ACE2) Receptor Binding Inhibition Assay Expressed as GMTs - Phase 1 | 189 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMTs at multiple time points through Day 189.
ACE2 Receptor Binding Inhibition Assay Expressed as GMFRs - Phase 1 | 189 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMFRs at multiple time points through Day 189.
ACE2 Receptor Binding Inhibition Assay Expressed as SCRs - Phase 1 | 189 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SCRs at multiple time points through Day 189.
ACE2 Receptor Binding Inhibition Assay Expressed as SRRs - Phase 1 | 189 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SRRs at multiple time points through Day 189.
Neutralizing Antibody Activity Expressed as GMTs - Phase 1 | 49 days
  Neutralizing antibody activity as detected by microneutralization assay (MN) expressed as GMTs at multiple time points through Day 49.
Neutralizing Antibody Activity Expressed as GMFRs - Phase 1 | 49 days
  Neutralizing antibody activity as detected by MN expressed as GMFRs at multiple time points through Day 49.
Neutralizing Antibody Activity Expressed as SCRs - Phase 1 | 49 days
  Neutralizing antibody activity as detected by MN expressed as SCRs at multiple time points through Day 49.
Neutralizing Antibody Activity Expressed as SRRs - Phase 1 | 49 days
  Neutralizing antibody activity as detected by MN expressed as SRRs at multiple time points through Day 49.
Assessment of Cell-Mediated (T helper 1 [Th1]/T helper 2 [Th2]) Pathways - Phase 1 | 28 days
  Cell-mediated (Th1/Th2) pathways as measured by whole blood (flow cytometry) and/or in vitro peripheral blood mononuclear cell (PBMC) stimulation (eg, enzyme-linked immunospot [ELISpot], cytokine staining) with SARS-CoV-2 rS protein(s) through Day 28.
Assessment of Serum IgG Antibody Levels Expressed as GMTs - Phase 2 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs for the single-dose regimens compared to the two-dose regimens and to placebo through Day 35 regardless of baseline immune status and stratified by baseline immune status.
Assessment of Serum IgG Antibody Levels Expressed as GMFRs - Phase 2 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs for the single-dose regimens compared to the two-dose regimens and to placebo through Day 35 regardless of baseline immune status and stratified by baseline immune status.
Assessment of Serum IgG Antibody Levels Expressed as SCRs (≥ 4-fold change) - Phase 2 | 35 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs (≥ 4-fold change) for the single-dose regimens compared to the two-dose regimens and to placebo through Day 35 regardless of baseline immune status and stratified by baseline immune status.
Assessment of Serum IgG Antibody Levels Expressed as GMEUs at Multiple Time Points - Phase 2 | 357 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo, stratified by baseline immune response.
Assessment of Serum IgG Antibody Levels Expressed as GMFRs at Multiple Time Points - Phase 2 | 357 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo, stratified by baseline immune response.
Assessment of Serum IgG Antibody Levels Expressed as SCRs (≥ 4-fold change) at Multiple Time Points - Phase 2 | 357 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as SCRs (≥ 4-fold change) at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo, stratified by baseline immune response.
ACE2 Receptor Binding Inhibition Assay Expressed as GMTs - Phase 2 | 357 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMTs at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo.
ACE2 Receptor Binding Inhibition Assay Expressed as GMFRs - Phase 2 | 357 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as GMFRs at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo.
ACE2 Receptor Binding Inhibition Assay Expressed as SCRs - Phase 2 | 357 days
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by ACE2 receptor binding inhibition assay expressed as SCRs (≥ 4-fold change) at multiple time points through Day 357 for the single-dose regimens compared to the two-dose regimens and to placebo.
Neutralizing Antibody Activity Expressed as GMTs - Phase 2 | 357 days
  Neutralizing antibody activity as detected by MN expressed as GMTs at Days 35, 217, and 357 relative to baseline in a subset of subjects by absolute titers and change from baseline.
Neutralizing Antibody Activity Expressed as GMFRs - Phase 2 | 357 days
  Neutralizing antibody activity as detected by MN expressed as GMFRs at Days 35, 217 and 357 relative to baseline in a subset of subjects by absolute titers and change from baseline.
Neutralizing Antibody Activity Expressed as SCRs (≥ 4-fold change) - Phase 2 | 357 days
  Neutralizing antibody activity as detected by MN expressed as SCRs (≥ 4-fold change) at Days 35, 217, and 357 relative to baseline in a subset of subjects by absolute titers and change from baseline.
Assessment of Serum IgG Antibody Levels Expressed as GMTs - Phase 2 Boost | 546 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at Days 189, 217, and 357 for all treatment groups and additionally at Day 371 and Day 546 for treatment groups B and C for boosting assessment with either placebo or active boost.
Assessment of Serum IgG Antibody Levels Expressed as GMFRs - Phase 2 Boost | 546 days
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Days 189, 217, and 357 for all treatment groups and additionally at Day 371 and Day 546 for treatment groups B and C for boosting assessment with either placebo or active boost.
Participants with MAAEs - Phase 2 | 217 days
  All MAAEs, defined as AEs that lead to an unscheduled visit to a healthcare practitioner, through Day 217 by MedDRA classification, severity score, and relatedness.
Participants with Related MAAEs; SAEs; and AESIs - Phase 2 | 357 days
  Percentage of participants with MAAEs assessed as related to study vaccine, SAEs, and AESIs until the end of the study (EOS) by MedDRA classification and severity score. All SAEs and AESI, defined as potential immune-mediated medical conditions or AEs relevant to COVID-19, by MedDRA classification, severity score, and relatedness.
Participants with Abnormal Vital Signs - Phase 2 | 21 days
  Percentage of participants with vital sign abnormalities on the day of vaccination by severity scoring immediately following vaccination. Descriptive statistics (mean, standard deviation, change from baseline) by treatment group, by visit.
Changes from Baseline in Body Temperature - Phase 2 | 189 days
  Mean changes from baseline in body temperature by treatment group and visit.
Changes from Baseline in Blood Pressure - Phase 2 | 189 days
  Mean changes from baseline in blood pressure by treatment group and visit.
Changes from Baseline in Pulse Rate - Phase 2 | 189 days
  Mean changes from baseline in pulse rate by treatment group and visit.
Participants with SARS-CoV-2 Positivity - Phase 2 | 161 days
  Percentage of participants with SARS-CoV-2 positivity as diagnosed by qualitative polymerase chain reaction (PCR) following COVID-19 symptoms assessment from Day 28 through 6 months with severity classification, overall and by age strata (18-59, 60-84 years).
Assessment of SARS-CoV-2 by Qualitative PCR - Phase 2 | 161 days
  Assessment of SARS-CoV-2 by qualitative PCR based on routine screening by self- collection (nasal mid-turbinate or saliva) from Day 28 through 6 months without symptomatology to further describe epidemiologic evolution of the pandemic and potential effect of vaccination.
Assessment of Cell-Mediated (Th1/Th2) Pathways - Phase 2 | 28 days
  Assessment of cell-mediated (Th1/Th2) pathways as measured by whole blood (flow cytometry) and/or in vitro PBMC stimulation (eg, ELISpot, cytokine staining) with SARS-CoV-2 rS protein(s) through Day 28.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (18):
- United States (8):
  - Meridian Clinical Research-(Savannah Georgia) - Platinum - PPDS - Phase 2, Savannah, Georgia
  - Advanced Clinical Research - Meridian - ERN-PPDS - Phase 2, Meridian, Idaho
  - Alliance for Multispecialty Research, LLC - Phase 2, Newton, Kansas
  - Alliance for Multispecialty Research, LLC - Phase 2, Wichita, Kansas
  - Central Kentucky Research Associates Inc - Phase 2, Lexington, Kentucky
  - Meridian Clinical Research-(Rockville Maryland) - Platinum - PPDS - Phase 2, Rockville, Maryland
  - Synexus Clinical Research US, Inc. - Cincinnati - Phase 2, Cincinnati, Ohio
  - Rapid Medical Research Inc - ERN-PPDS - Phase 2, Cleveland, Ohio
- Australia (10):
  - Paratus Clinical Research - Canberra - Phase 2, Bruce, Australian Capital Territory
  - Paratus Clinical Research - Western Sydney - Phase 2, Blacktown, New South Wales
  - Paratus Clinical Research - Central Coast - Phase 2, Kanwal, New South Wales
  - Australian Clinical Research Network - Phase 2, Maroubra, New South Wales
  - Scientia Clinical Research Limited - Phase 2, Randwick, New South Wales
  - Q Pharm Pty Limited - Phase 1, Herston, Queensland
  - University of the Sunshine Coast, Health Hub Morayfield - Phase 2, Morayfield, Queensland
  - University of the Sunshine Coast - Phase 2, Sippy Downs, Queensland
  - Barwon Health - Phase 2, Geelong, Victoria
  - Center for Clinical Studies - Phase 1 and Phase 2, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bangaru S, Jackson AM, Copps J, Fernandez-Quintero ML, Torres JL, Richey ST, Nogal B, Sewall LM, Torrents de la Pena A, Rehman A, Guebre-Xabier M, Girard B, Das R, Corbett-Helaire KS, Seder RA, Graham BS, Edwards DK, Patel N, Smith G, Ward AB. Structural serology of polyclonal antibody responses to mRNA-1273 and NVX-CoV2373 COVID-19 vaccines. Cell Rep. 2025 Jul 22;44(7):115986. doi: 10.1016/j.celrep.2025.115986. Epub 2025 Jul 8. PMID 40632654
- [Derived] Alves K, Plested JS, Galbiati S, Chau G, Cloney-Clark S, Zhu M, Kalkeri R, Patel N, Smith K, Marcheschi A, Pfeiffer S, McFall H, Smith G, Glenn GM, Dubovsky F, Mallory RM; Novavax 2019nCoV-101 Study Group. Immunogenicity and safety of a fourth homologous dose of NVX-CoV2373. Vaccine. 2023 Jun 29;41(29):4280-4286. doi: 10.1016/j.vaccine.2023.05.051. Epub 2023 Jun 2. PMID 37271706
- [Derived] Fries L, Formica N, Mallory RM, Zhou H, Plested JS, Kalkeri R, Moldovan I, Patel N, Albert G, Robinson M, Cho I, Chau G, Dubovsky F, Glenn GM; 2019nCoV-101 Study Group. Strong CD4+ T-Cell Responses to Ancestral and Variant Spike Proteins Are Established by NVX-CoV2373 Severe Acute Respiratory Syndrome Coronavirus 2 Primary Vaccination. J Infect Dis. 2023 Sep 15;228(6):734-741. doi: 10.1093/infdis/jiad163. PMID 37210741
- [Derived] Mallory RM, Formica N, Pfeiffer S, Wilkinson B, Marcheschi A, Albert G, McFall H, Robinson M, Plested JS, Zhu M, Cloney-Clark S, Zhou B, Chau G, Robertson A, Maciejewski S, Hammond HL, Baracco L, Logue J, Frieman MB, Smith G, Patel N, Glenn GM; Novavax 2019nCoV101 Study Group. Safety and immunogenicity following a homologous booster dose of a SARS-CoV-2 recombinant spike protein vaccine (NVX-CoV2373): a secondary analysis of a randomised, placebo-controlled, phase 2 trial. Lancet Infect Dis. 2022 Nov;22(11):1565-1576. doi: 10.1016/S1473-3099(22)00420-0. Epub 2022 Aug 10. PMID 35963274
- [Derived] Formica N, Mallory R, Albert G, Robinson M, Plested JS, Cho I, Robertson A, Dubovsky F, Glenn GM; 2019nCoV-101 Study Group. Different dose regimens of a SARS-CoV-2 recombinant spike protein vaccine (NVX-CoV2373) in younger and older adults: A phase 2 randomized placebo-controlled trial. PLoS Med. 2021 Oct 1;18(10):e1003769. doi: 10.1371/journal.pmed.1003769. eCollection 2021 Oct. PMID 34597298
- [Derived] Tian JH, Patel N, Haupt R, Zhou H, Weston S, Hammond H, Logue J, Portnoff AD, Norton J, Guebre-Xabier M, Zhou B, Jacobson K, Maciejewski S, Khatoon R, Wisniewska M, Moffitt W, Kluepfel-Stahl S, Ekechukwu B, Papin J, Boddapati S, Jason Wong C, Piedra PA, Frieman MB, Massare MJ, Fries L, Bengtsson KL, Stertman L, Ellingsworth L, Glenn G, Smith G. SARS-CoV-2 spike glycoprotein vaccine candidate NVX-CoV2373 immunogenicity in baboons and protection in mice. Nat Commun. 2021 Jan 14;12(1):372. doi: 10.1038/s41467-020-20653-8. PMID 33446655
- [Derived] Guebre-Xabier M, Patel N, Tian JH, Zhou B, Maciejewski S, Lam K, Portnoff AD, Massare MJ, Frieman MB, Piedra PA, Ellingsworth L, Glenn G, Smith G. NVX-CoV2373 vaccine protects cynomolgus macaque upper and lower airways against SARS-CoV-2 challenge. Vaccine. 2020 Nov 25;38(50):7892-7896. doi: 10.1016/j.vaccine.2020.10.064. Epub 2020 Oct 23. PMID 33139139
- [Derived] Keech C, Albert G, Cho I, Robertson A, Reed P, Neal S, Plested JS, Zhu M, Cloney-Clark S, Zhou H, Smith G, Patel N, Frieman MB, Haupt RE, Logue J, McGrath M, Weston S, Piedra PA, Desai C, Callahan K, Lewis M, Price-Abbott P, Formica N, Shinde V, Fries L, Lickliter JD, Griffin P, Wilkinson B, Glenn GM. Phase 1-2 Trial of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine. N Engl J Med. 2020 Dec 10;383(24):2320-2332. doi: 10.1056/NEJMoa2026920. Epub 2020 Sep 2. PMID 32877576